CLINICAL TRIAL: NCT01714050
Title: Cognitive-behavioral Therapy vs. Light Therapy for Preventing Seasonal Affective Disorder Recurrence
Brief Title: Cognitive-behavioral Therapy vs. Light Therapy for Preventing SAD Recurrence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kelly Rohan, Associate Professor of Psychology, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: R01MH078982 (NIH); R01MH078982 (NIH)
Record Dates: First submitted 2012-10-17; First posted 2012-10-25 (Estimated); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Seasonal Affective Disorder (SAD); Winter Depression; Major Depressive Disorder, Recurrent, With Seasonal Pattern
Keywords: seasonal affective disorder; winter depression; cognitive-behavioral therapy; light therapy
MeSH Terms: conditions — Seasonal Affective Disorder; Depressive Disorder, Major; Recurrence | interventions — Cognitive Behavioral Therapy; Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cognitive-Behavioral Therapy (CBT) (Experimental): The CBT is a SAD-tailored version of Beck et al.'s (1979) cognitive therapy for depression called "Coping with the Seasons" (Rohan, 2008). The rationale addresses environmental changes, thoughts, and behaviors in SAD onset and maintenance. It seeks to change behaviors and thoughts to improve coping with winter. Behaviors that promote enjoyment in the winter are increased. Negative thoughts that interfere with self-esteem and negative thoughts about winter are identified and addressed. A relapse-prevention component addresses early identification of negative anticipatory thoughts about winter and SAD-related behavior changes, using the CBT skills learned to cope with subsequent winter seasons, and development of a personalized relapse-prevention plan. The CBT sessions are administered twice a week over 6 weeks (total of 12 sessions) with 4-8 participants per group. The CBT is led by one of three licensed Ph.D.-level psychologists working on the project.
  Interventions: Behavioral: Cognitive-Behavioral Therapy (CBT)
- Light Therapy (LT) (Experimental): LT will be initiated at 30-minutes in the morning at home, first thing upon awakening, using a light box with an ultraviolet shield that emits 10,000-lux of white fluorescent light. After the first week, an M.D. light therapy consultant will recommend individually-tailored, clinical adjustments to the duration and timing of light use to maximize response and reduce any reported side effects. For each of the 6-weeks of LT, LT participants will complete a Light Therapy Side Effects Questionnaire to assess side effects attributed to LT. Participants will keep daily LT compliance diaries to record the timing and duration of LT. After the 6-weeks of monitoring, participants may choose to continue using the light box through April. We will offer LT participants who wish to use light therapy in the next fall/winter season access to our light boxes if they agree to followup with a physician or other qualified professional for monitoring and side effects management.
  Interventions: Device: Light Therapy (LT)

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy (CBT)
  Arms: Cognitive-Behavioral Therapy (CBT)
Device: Light Therapy (LT) — SunRay (SunBox Company, Gaithersburg, MD)
  Arms: Light Therapy (LT)

SUMMARY:
Major depression is a highly prevalent, chronic, and debilitating mental health problem with significant social cost that poses a tremendous economic burden. Winter seasonal affective disorder (SAD) is a subtype of recurrent major depression involving substantial depressive symptoms that adversely affect the family and workplace for about 5 months of each year during most years, beginning in young adulthood. This clinical trial is relevant to this public health challenge in seeking to develop and test a time-limited (i.e., acute treatment completed in a discrete period vs. daily treatment every fall/winter indefinitely), palatable cognitive-behavioral treatment with effects that endure beyond the cessation of acute treatment to prevent the annual recurrence of depression in SAD.

Aim (1) To compare the long-term efficacy of cognitive-behavioral therapy (CBT) and light therapy on depression recurrence status, symptom severity, and remission status during the next winter season (i.e., the next wholly new winter season after the initial winter of treatment completion), which we argue to be the most important time point for evaluating clinical outcomes following SAD intervention.

Hypothesis: CBT will be associated with a smaller proportion of depression recurrences, less severe symptoms, and a higher proportion of remissions than light therapy in the next winter. The study is designed to detect a clinically important difference between CBT and light therapy in depressive episode recurrences during the next winter, the primary endpoint, in an intent-to-treat analysis.

Aim (2) To compare the efficacy of CBT and light therapy on symptom severity and remission status at post-treatment (treatment endpoint).

Hypothesis: CBT and light therapy will not differ significantly on post-treatment outcomes.

DETAILED DESCRIPTION:
Seasonal affective disorder (SAD) is a subtype of recurrent depression involving major depressive episodes during the fall and/or winter months that remit in the spring. SAD affects an estimated 5% of the U. S. population, over 14.5 million Americans. The central public health challenge in the management of SAD is prevention of winter depression recurrence. The established and best available treatment, light therapy, remits acute symptoms in 53% of SAD cases. However, long-term compliance with clinical practice guidelines recommending daily use of a light box from onset of first symptom through spontaneous springtime remission during every fall/winter season is poor. Time-limited alternative treatments with durable effects are needed to prevent the annual recurrence of these disabling symptoms. Our preliminary studies suggest that a novel, SAD-tailored cognitive-behavioral therapy (CBT) may be as efficacious as light therapy alone for acute SAD treatment and that CBT may have superior outcomes to light therapy during the next winter. During the next wholly new winter season following the initial winter of study treatment, the proportion of depression recurrences was significantly smaller in participants randomized to CBT (5.8%) or to CBT combined with light therapy (5.2%) than in participants randomized to light therapy alone (39.2%). As the next step in this programmatic line of intervention studies, the primary aim of the proposed project is to further test the efficacy of our CBT for SAD intervention against light therapy in a larger, more definitive randomized head-to-head comparison on next winter outcomes in an intent-to-treat (ITT) analysis using all randomized participants. This project is seeking to test for a clinically meaningful difference between CBT and light therapy on depression recurrence in the next winter (the primary outcome), thereby having the potential to impact clinical practice. The proposed work will go beyond our pilot studies in four ways: (1) This study will augment the generalizability of our prior pilot study data by relaxing the inclusion/exclusion criteria to allow for comorbid diagnoses and stable antidepressant medication use and by demonstrating the feasibility of training experienced community therapists to facilitate the CBT groups. (2) We will prospectively track recurrences and potential intervening variables that could affect outcome (e.g., new treatments, summer remission status) in the interim between treatment endpoint and the following winter. (3) This study includes a second annual winter followup to obtain preliminary data on the comparative effects of CBT vs. LT two winters after the initial winter of study treatment. (4) We will examine how potential modifiers influence the effects of CBT vs. LT, including demographic variables; baseline characteristics (e.g., depression severity, comorbidity, baseline medication status); and complete or incomplete summer remission status in the interim. If successful, this work will develop a novel treatment with important public health implications for winter depression prevention.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 or older
* meet DSM-IV criteria for Major Depression, Recurrent, with Seasonal Pattern
* meet Structured Interview Guide for the Hamilton Rating Scale for Depression-Seasonal Affective Disorder Version (SIGH-SAD) criteria for a current SAD episode

Exclusion Criteria:

* past light therapy or cognitive-behavioral therapy for SAD
* presence of a comorbid Axis I disorder that requires immediate treatment
* acute and serious suicidal intent
* positive laboratory findings for hypothyroidism
* plans for major vacations or absences from the study area through March

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2008-07; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Depression recurrence status on the Structured Interview Guide for the Hamilton Rating Scale for Depression-Seasonal Affective Disorder Version (SIGH-SAD; Williams et al., 1992) | next winter followup (January or February of the next winter, approximately a year after study treatment)
  The SIGH-SAD (Williams et al., 1992), the most commonly used clinical assessment device for detecting changes in SAD symptoms in light therapy research, includes the 21-item Structured Interview Guide for the Hamilton Rating Scale for Depression (HAM-D) and a supplementary 8-item subscale to assess atypical depressive symptoms associated with SAD. The primary outcome measure is SIGH-SAD recurrence status at the next winter followup. A trained rater, blind to the treatment condition, will administer the SIGH-SAD at pre-treatment, treatment weeks 1-5, post-treatment, summer followup, next winter followup, and second winter followup. A second blinded rater will rate audiotapes of the SIGH-SADs to assess inter-rater reliability.

SECONDARY OUTCOMES:
Beck Depression Inventory-Second Edition (BDI-II; Beck et al., 1996) | baseline, mid-treatment (week 3), post-treatment (week 6), summer followup (August), next winter followup (January or February or the next winter), and the second winter followup (January or February two winters later)
  The BDI-II (Beck et al., 1996) is a 21-item measure of depressive symptom severity. The BDI-II has demonstrated good test-retest reliability and convergent validity (Beck et al., 1996). This study will use the BDI-II as a continuous measure of depressive symptom severity. Studies have also used the BDI-II to estimate remission rates subsequent to treatment (Gortner et al., 1996). Therefore, dichomotous remission status on the BDI-II will also be assessed. The BDI-II will be administered at baseline, mid-treatment (week 3) and post-treatment (week 6), summer followup, next winter followup, and the second winter followup.
Structured Interview Guide for the Hamilton Rating Scale for Depression-Seasonal Affective Disorder Version (SIGH-SAD) | baseline, weekly during treatment (weeks 1-5), post-treatment (week 6), summer followup (August), next winter followup (January or February of the next winter), second winter followup (January or February two winters later)
  In addition to the primary outcome of SIGH-SAD depression recurrence status, other secondary measures based on the SIGH-SAD will include continuous SIGH-SAD scores and SIGH-SAD remission status.

CONTACTS AND LOCATIONS:
Overall Officials: Kelly J Rohan, Ph.D., Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Psychology Department, Burlington, Vermont, United States

REFERENCES:
- [Derived] Rohan KJ, Terman JM, Iyiewuare P, Perez J, Camuso JA, Postolache TT, DeSarno MJ, Vacek PM. Prospectively assessed summer mood status in major depression, recurrent with seasonal pattern: Evidence for SAD's construct validity. J Affect Disord. 2024 Mar 15;349:32-38. doi: 10.1016/j.jad.2023.12.070. Epub 2023 Dec 30. PMID 38160889
- [Derived] Rohan KJ, Burt KB, Norton RJ, Perez J, Iyiewuare P, Terman JM. Change in Seasonal Beliefs Mediates the Durability Advantage of Cognitive-Behavioral Therapy Over Light Therapy for Winter Depression. Behav Ther. 2023 Jul;54(4):682-695. doi: 10.1016/j.beth.2022.11.002. Epub 2022 Dec 7. PMID 37330257
- [Derived] Terman JM, Rohan KJ, Stickle TR, Wernhoff A. Personality Pathology in Winter Depression: Prevalence and Treatment Trajectories in Cognitive-Behavioral Therapy and Light Therapy. Behav Ther. 2023 Mar;54(2):361-374. doi: 10.1016/j.beth.2022.10.002. Epub 2022 Nov 2. PMID 36858765
- [Derived] Rohan KJ, Burt KB, Camuso J, Perez J, Meyerhoff J. Applying experimental therapeutics to examine cognitive and chronological vulnerabilities as mediators of acute outcomes in cognitive-behavioral therapy and light therapy for winter depression. J Consult Clin Psychol. 2020 Aug;88(8):786-797. doi: 10.1037/ccp0000499. PMID 32700956
- [Derived] Rohan KJ, Meyerhoff J, Ho SY, Evans M, Postolache TT, Vacek PM. Outcomes One and Two Winters Following Cognitive-Behavioral Therapy or Light Therapy for Seasonal Affective Disorder. Am J Psychiatry. 2016 Mar 1;173(3):244-51. doi: 10.1176/appi.ajp.2015.15060773. Epub 2015 Nov 5. PMID 26539881
- [Derived] Rohan KJ, Mahon JN, Evans M, Ho SY, Meyerhoff J, Postolache TT, Vacek PM. Randomized Trial of Cognitive-Behavioral Therapy Versus Light Therapy for Seasonal Affective Disorder: Acute Outcomes. Am J Psychiatry. 2015 Sep 1;172(9):862-9. doi: 10.1176/appi.ajp.2015.14101293. Epub 2015 Apr 10. PMID 25859764
- [Derived] Rohan KJ, Evans M, Mahon JN, Sitnikov L, Ho SY, Nillni YI, Postolache TT, Vacek PM. Cognitive-behavioral therapy vs. light therapy for preventing winter depression recurrence: study protocol for a randomized controlled trial. Trials. 2013 Mar 21;14:82. doi: 10.1186/1745-6215-14-82. PMID 23514124